CLINICAL TRIAL: NCT05816057
Title: A Multicenter, Randomized, Open-label, and Parallel Assignment Phase III Study to Compare the Efficacy and Safety of Semaglutide Injection With Ozempic® in Combination With Metformin in the Treatment of Type 2 Diabetes
Brief Title: A Study of the Efficacy and Safety of Semaglutide Injection in the Treatment of Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Jiuyuan Gene Engineering Co. Ltd., (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JY-2021-05
Record Dates: First submitted 2023-02-20; First posted 2023-04-18 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- semaglutide injection (Experimental): Semaglutide 0.25 mg、0.5 mg、1.0mg
  Interventions: Biological: semaglutide injection
- ozempic® (Active Comparator): Ozempic® 0.25 mg、0.5 mg、1.0mg
  Interventions: Biological: semaglutide injection

INTERVENTIONS:
Biological: semaglutide injection — The subject will receive either a dose semaglutide once weekly (subcutaneous (s.c.) injection). The initial dose of 0.25 mg is s.c. once weekly, and the dose is increased to 0.5 mg after 4 weeks of administration, and the dose is increased to 1 mg after 4 weeks of 0.5 mg administration, and the dose is continued at a stable dose of 1 mg for 24 weeks.Treatment duration 32 weeks.

SUMMARY:
Semaglutide injection is a new drug developed according to Ozempic® biosimilars.This trial is conducted in China. The purpose of this study is to investigate the similarities in the efficacy and safety of semaglutide injection and Ozempic® in the treatment of type 2 diabetes, respectively.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, open-label, parallel assignment, which plans to enroll 476 patients with type 2 diabetes And Stable daily dose for 4 weeks prior to the day of screening of the metformin formulations (greater than or equal to 1500 mg to less than or equal to 2000 mg or maximum tolerated dose documented greater than or equal to 1000 mg. The study was divided into three phases: screening, baseline and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in the trial and sign the informed consent form；
2. Diagnosed with type 2 diabetes And Stable daily dose for 4 weeks prior to the day of screening of the metformin formulations (greater than or equal to 1500 mg to less than or equal to 2000 mg or maximum tolerated dose documented greater than or equal to 1000 mg)；
3. Male or female, Aged 18-75 years (both inclusive) at the time of signing informed consent；
4. Glycated haemoglobin (HbA1c) of greater than 7.0% to less than or less than or equal to 11.0%.

Exclusion Criteria:

1. Treatment with any medication for the indication of diabetes other than stated in the inclusion criteria within the past 4 weeks prior to the day of screening. However, short-term insulin treatment for a maximum of 7 days prior to the day of screening is allowed;
2. Systemic corticosteroids (excluding topical and inhaled preparations) within the past 90 days to the day of screening;
3. Known or suspected hypersensitivity to trial product(s) or related products;
4. Have participated in other clinical trials and used investigational drugs within the past 90 days to the day of screening;
5. Heart failure(Subjects presently classified as being in New York Heart Association Class IV); Acute coronary syndrome or cerebrovascular events, including but not limited to acute myocardial infarction, stroke, unstable angina or transient ischaemic attack; Have undergone heart-related surgery; or investigator assessment of severe ECG abnormalities, poorly controlled hypertension (defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg), and other cardiovascular and cerebrovascular disorders that are not suitable within the past 90 days prior to the day of screening;
6. Known to plan to be hospitalized for any surgery at the time of screening;
7. Hyperthyroidism, Cushing's syndrome, Diabetic gastroparesis or other gastrointestinal disorders; Gastrointestinal disorders assessed by investigators as increasing post-medication risk, anorexia, alcohol dependence, drug use, drug dependence, epilepsy, psychiatric illness, need for systemic anti-infective therapy, or other conditions assessed by investigators as affecting endpoint assessment;
8. Family or personal history of Multiple Endocrine Neoplasia Type 2 (MEN 2) or Medullary Thyroid Carcinoma (MTC);
9. History or presence of pancreatitis (acute or chronic);
10. Proliferative diabetic retinopathy.
11. Recurrent severe hypoglycaemia (more than 3 severe hypoglycaemic events) within the past 90 days to the day of screening;
12. Acute metabolic complications within the past 180 days prior to the day of screening;
13. Subjects with calcitonin ≥ 50 ng/L pg/mL) ,AMY ≥3×upper normal limit (UNL), triglyceride ≥5.7 mmol/L( 500 mg/dL) ,eGFR<60 mL/min/1.73 m2,; hemoglobin ≤120 g/L (male) or ≤110 g/L (female), ALT、AST≥ 2.5 ×UNL,TBIL≥2×ULN;
14. History or presence of malignant neoplasms within the last 5 years (except basal or squamous cell skin cancer and carcinoma in situ);
15. The female who is pregnant, breast-feeding or Female/male intends to become pregnant or is of child-bearing potential and not using highly effective contraceptive method; （16））Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2022-07-25 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
The observed mean change in Glycosylated Haemoglobin A1c (HbA1c) values from baseline after 32 weeks of treatment. | 32 weeks

SECONDARY OUTCOMES:
The observed mean change in HbA1c values from baseline after 20 weeks of treatment. | 20 weeks
Change From Baseline to Week 20 in Fasting Plasma Glucose (FPG). | 20 weeks
Change From Baseline to Week 32 in Fasting Plasma Glucose (FPG). | 32 weeks
Change From Baseline to Week 32 in HbA1c < 7.0% of participants. | 32 weeks
Change From Baseline to Week 32 in HbA1c≤6.5% of participants. | 32 weeks
Change From Baseline to Week 32 in HbA1c < 7.0% of participants with no hypoglycemic events. | 32 weeks
Change From Baseline to Week 32 in Body Weight (Kilogram (kg)). | 32 weeks
Change From Baseline to Week 32 in Systolic and Diastolic Blood Pressure. | 32 weeks
Change From Baseline to Week 32 in Pulse Rate. | 32 weeks
Change From Baseline to Week 32 in Fasting Blood Lipids: Total Cholesterol、Low-density Lipoprotein (LDL) Cholesterol、 High-density Lipoprotein (HDL) Cholesterol 、Triglycerides (Ratio to Baseline). | 32weeks

CONTACTS AND LOCATIONS:
Overall Officials: xiaoying Li, M.D., Principal Investigator — Shanghai Zhongshan Hospital
Locations (35):
- China (35):
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - NanFang Hospital, Guangzhou, Guangdong
  - CANGZHOU People's Hospital, Cangzhou, Hebei
  - CANGZHOU Central Hospital, Cangzhou, Hebei
  - Cang zhou Hospital of Integrated Traditional Chinese and Western of Hebei Province, Cangzhou, Hebei
  - Shijiazhuang Second Hospital, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Nanyang First People's Hospital, Nanyang, Henan
  - Nanyang Second General Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Huangshi Central Hospital, Huangshi, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - Huizhou Central People's Hospital, Guangdong, Huizhou
  - Yueyang People's Hospital, Yueyang, Hunan
  - BaogangHospital of InnerMongolia, Baotou, Inner Mongolia
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - Huai'an Second People's Hospital, Huaian, Jiangsu
  - The Affiliated Huaian No.1 People's Hospital of Nanjing Medical University, Huaian, Jiangsu
  - The Second People's Hospital of Lianyungang, Lianyungang, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital OF Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xuzhou Cancer Hospital, Xuzhou, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhengjiang, Jiangsu
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - The First Affiliated Hospital of Xi'an jiaotong university, Xi'an, Shaanxi
  - Central Hospital Affiliated to Shandong First Medical University, Jinan, Shandong
  - Huadong Hospital Affillated to Fudan University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pudong New Area People's Hospital, Shanghai, Shanghai Municipality
  - Jincheng Grand Hospital, Jincheng, Shanxi
  - Shanxi Yuncheng Central Hospital, Yuncheng, Shanxi
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No